CLINICAL TRIAL: NCT02165540
Title: The Impact of Doulas in the Surgical Management of Early Pregnancy Failure and Abortion Care
Brief Title: The Impact of Doulas in Early Pregnancy Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Courtney Schreiber, Assistant Professor, Obstetrics and Gynecology, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 819173
Record Dates: First submitted 2014-05-19; First posted 2014-06-17 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Uterine Evacuation
Keywords: Doula; Pain management; Miscarriage; Abortion
MeSH Terms: conditions — Agnosia; Abortion, Spontaneous | interventions — Doulas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Doula (Experimental): Patients will have a doula support person during their procedure.
  Interventions: Other: Doula
- Routine care/No Doula (No Intervention): Patients will have routine care with clinical staff only.

INTERVENTIONS:
Other: Doula — A specially trained support person or doula will accompany the patient to offer physical and emotional support during the procedure.
  Arms: Doula

SUMMARY:
The purpose of the study is to examine the impact of doula support for women undergoing a manual vacuum aspiration (MVA) for an early pregnancy failure or undesired pregnancy.

DETAILED DESCRIPTION:
As a means of providing emotional support and physical comfort for all pregnant women, doulas have emerged in recent years in the world of clinical abortion care. Traditionally, doulas are non-medical individuals trained to provide emotional support, pain management strategies, relaxation techniques, and information to pregnant women during labor. The positive impact of doulas on obstetrical health outcomes and patient satisfaction is well accepted.

Women with the support of a doula have been shown to have shorter labor, and rate birth as less difficult and more satisfying, than do mothers without doula support. They also report a greater ability to cope with labor and require less epidural and IV pain medication. In recent years, the term full spectrum doula has emerged to describe doulas who extend their supportive services to women at any stage of a pregnancy, including the management of a miscarriage or undesired pregnancy ending in abortion. The Doula Project, created in 2007 in New York City, and the Bay Area Doula Project, founded in 2011in San Francisco, were two of the first organized efforts to train doulas to provide abortion care and are now the largest in the United States. Scientific research on the impact of doulas during abortion and miscarriage management has been limited, but anecdotal reports from patients and providers suggest a positive impact on patient satisfaction. In this study we aim to test the impact of doulas on the physical, emotional, and overall experience among women undergoing a MVA for an early pregnancy failure or undesired pregnancy at the Penn Family Planning and Pregnancy Loss Center. We also aim to assess the impact of doula support from the medical assistants perception.

ELIGIBILITY:
Inclusion Criteria:

* Female 18 years or older who is choosing to have a surgical procedure for the management of early pregnancy failure or undesired pregnancy.
* Pregnancy is not because of an incident of sexual assault or rape.

Exclusion Criteria:

* Pregnancy is due to an incident of sexual assault or rape.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The degree of physical discomfort reported by women during their MVA procedure. | At enrollment baseline
  This data is obtained in-clinic via a brief questionnaire after the patient undergoes the MVA at enrollment baseline.

SECONDARY OUTCOMES:
The degree to which women report the ability to emotionally cope with their MVA procedure. | At baseline visit and at 1-month follow-up
  This data was obtained via a brief questionnaire before and after the MVA at enrollment baseline, and then via a brief survey completed over the phone 1 month after enrollment.
The degree to which women sense empowerment before and following their MVA procedure | At enrollment baseline and 1-month follow-up
  This data was obtained via a brief questionnaire before and after the MVA at enrollment baseline, and then via a brief survey completed over the phone 1 month after enrollment.
A rating of the emotional response experienced by women before and after their MVA procedure. | At enrollment baseline and 1-month follow up
  This data was obtained via a brief questionnaire before and after the MVA at enrollment baseline, and then via a brief survey completed over the phone 1 month after enrollment.
The degree to which women are satisfied by their MVA procedure experience | At enrollment baseline and 1-month follow-up
  This data was obtained via a brief questionnaire after the MVA at enrollment baseline, and then via a brief survey completed over the phone 1 month after enrollment.
The degree to which medical assistant reports a more positive or negative patient and personal experience with the MVA procedure | At enrollment baseline
  This data will be obtained via a Visual Analog Scale administered after the MVA procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Schreiber, MD, MPH, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Family Planning and Pregnancy Loss Center, Philadelphia, Pennsylvania, United States